CLINICAL TRIAL: NCT05144152
Title: A Prospective Study to Assess the Diagnostic Accuracy of a Panel of Bacterial Gene Markers (M3) in Predicting Colorectal Advanced Adenoma Recurrence
Brief Title: Diagnostic Accuracy of M3 in Predicting Colorectal Advanced Adenoma Recurrence (M3-AA)
Acronym: M3-AA
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Louis Ho Shing Lau, Resident Specialist, Chinese University of Hong Kong
Other Study IDs: 2021.558
Record Dates: First submitted 2021-11-21; First posted 2021-12-03 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Adenoma; Advanced Adenoma; Colorectal Polyp
Keywords: FIT; Bacterial marker; Colonoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- History of colorectal adenomas group: Subjects with known colorectal adenomas at the index colonoscopy
  Interventions: Diagnostic Test: M3; Diagnostic Test: FIT

INTERVENTIONS:
Diagnostic Test: M3 — A panel of four bacterial gene markers (Fn, m3, Ch and Bc)
Diagnostic Test: FIT — faecal immunochemical test

SUMMARY:
The investigators aim to evaluate the diagnostic accuracy of FIT and the novel panel of four bacterial gene markers collectively named as M3, to detect recurrent advanced adenomas in patients with history of colonic adenomas.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the most common cancer in Hong Kong with more than 5,600 new cases annually. There is prevailing evidence of increasing trend of young onset CRC globally. Early detection and endoscopic resection of pre-malignant colonic adenomas has shown to reduce CRC-related mortality.

After the index colonoscopy, a surveillance colonoscopy will be required at regular intervals, depending on the number, size and histology of colonic polyps. Studies have reported the use of faecal immunochemical test (FIT) to reduce the burden on surveillance endoscopy service. However, approximately 30-40% of interval CRC and 40-70% of advanced adenomas (AA) could be missed by this strategy. The major limitation of this widely used non-invasive stool test is its unsatisfactory sensitivities for CRC (79%) and AA (40%). The sensitivity for non-advanced adenomas is even lower than 10%. A large proportion of advanced and non-advanced adenomas will be missed by FIT alone. Therefore, identification of alternative non-invasive test with better sensitivity to detect colonic adenomas is warranted.

Multitarget stool DNA test and faecal microbial DNA markers appear to be the most promising stool-based diagnostic biomarkers for screening CRC. Several bacterial gene markers have been identified by metagenome sequencing and reported to be associated with CRC, including Fusobacterium nucleatum (Fn), Clostridium hathewayi (Ch) and Bacteroides clarus (Bc). However, these molecular markers had low accuracy in distinguishing adenomas from normal tissue. Recently, a new Lachnoclostridium gene marker (labelled as 'm3') has been shown to have high diagnostic yield for the detection of colorectal adenomas. In a case-control study of 1012 subjects, a linear increasing trend of m3 level was observed from fecal samples of healthy subjects to those with adenomas and cancers. The overall sensitivity of m3 was significantly higher than FIT in detecting all adenomas (48% vs 9.3%), AA (50.8% vs 16.1%) and non-advanced adenomas (44.2% vs 0%). The diagnostic accuracy of m3 could be further enhanced by combining with a panel of fecal microbial markers composing of Fusobacterium nucleatum (Fn), Bacteroides clarus (Bc), Clostridium hathewayi (Ch) for CRC (82.3%) and adenomas (64.2%). The combination of these 4 bacterial gene markers (known as M3) has recently been proven to be useful in detecting adenoma recurrence after polypectomy in a retrospective study. The hypothesis is that it would be effective in the detection of recurrent advanced adenomas.

This prospective cohort study aims to evaluate the diagnostic accuracy of FIT and the novel panel of four bacterial gene markers (Fn, m3, Ch and Bc) collectively named as M3, to detect recurrent advanced adenomas in patients with history of colonic adenomas.

ELIGIBILITY:
Inclusion Criteria:

1. Known colorectal adenomas during index colonoscopy;
2. Available baseline M3 and FIT results before index colonoscopy;
3. Aged ≥18 years old;
4. Written informed consent obtained.

Exclusion Criteria:

1. Refusal or unfit to undergo surveillance colonoscopy;
2. Incomplete colonoscopy, incomplete removal of colorectal adenomas, or inadequate bowel preparation (defined as Boston Bowel Preparation Scale score 0 or 1 in any colonic segment) at index colonoscopy;
3. Previous colonic resection;
4. Personal history of colorectal cancer;
5. Personal history of polyposis syndrome;
6. Personal history of inflammatory bowel disease;
7. Known pregnancy or lactation;
8. Advanced comorbid conditions (defined as American Society of Anesthesiologists grade 4 or above);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subeject with history of colorectal adenomas
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the panel of bacterial gene markers (M3) or FIT in detection of recurrent colonic advanced adenomas | 3 years
  The proportion of subjects with true positive results of either M3 or FIT among those with one of more advanced adenomas detected during the surveillance colonoscopy examination at year 3

SECONDARY OUTCOMES:
Sensitivity for advanced adenomas (year 3) | 3 years
  The proportion of subjects with true positive results of either M3 or FIT among those with one of more advanced adenomas detected at year 3 colonoscopy
Sensitivity for non-advanced adenomas (year 3) | 3 years
  The proportion of subjects with true positive results of either M3 or FIT among those with non-advanced adenomas detected at year 3 colonoscopy
Sensitivity for all adenomas (year 3) | 3 years
  The proportion of subjects with true positive results of either M3 or FIT among those with all adenomas detected at year 3 colonoscopy
Specificity (year 3) | 3 years
  Proportion of true negative results of M3/FIT among those with no adenoma detected in colonoscopy (year 3)

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data to other researchers

REFERENCES:
- [Background] Yu J, Feng Q, Wong SH, Zhang D, Liang QY, Qin Y, Tang L, Zhao H, Stenvang J, Li Y, Wang X, Xu X, Chen N, Wu WK, Al-Aama J, Nielsen HJ, Kiilerich P, Jensen BA, Yau TO, Lan Z, Jia H, Li J, Xiao L, Lam TY, Ng SC, Cheng AS, Wong VW, Chan FK, Xu X, Yang H, Madsen L, Datz C, Tilg H, Wang J, Brunner N, Kristiansen K, Arumugam M, Sung JJ, Wang J. Metagenomic analysis of faecal microbiome as a tool towards targeted non-invasive biomarkers for colorectal cancer. Gut. 2017 Jan;66(1):70-78. doi: 10.1136/gutjnl-2015-309800. Epub 2015 Sep 25. PMID 26408641
- [Background] Liang JQ, Wong SH, Szeto CH, Chu ES, Lau HC, Chen Y, Fang J, Yu J, Sung JJ. Fecal microbial DNA markers serve for screening colorectal neoplasm in asymptomatic subjects. J Gastroenterol Hepatol. 2021 Apr;36(4):1035-1043. doi: 10.1111/jgh.15171. Epub 2020 Jul 15. PMID 32633422
- [Background] Liang Q, Chiu J, Chen Y, Huang Y, Higashimori A, Fang J, Brim H, Ashktorab H, Ng SC, Ng SSM, Zheng S, Chan FKL, Sung JJY, Yu J. Fecal Bacteria Act as Novel Biomarkers for Noninvasive Diagnosis of Colorectal Cancer. Clin Cancer Res. 2017 Apr 15;23(8):2061-2070. doi: 10.1158/1078-0432.CCR-16-1599. Epub 2016 Oct 3. PMID 27697996
- [Background] Wong SH, Kwong TNY, Chow TC, Luk AKC, Dai RZW, Nakatsu G, Lam TYT, Zhang L, Wu JCY, Chan FKL, Ng SSM, Wong MCS, Ng SC, Wu WKK, Yu J, Sung JJY. Quantitation of faecal Fusobacterium improves faecal immunochemical test in detecting advanced colorectal neoplasia. Gut. 2017 Aug;66(8):1441-1448. doi: 10.1136/gutjnl-2016-312766. Epub 2016 Oct 24. PMID 27797940
- [Background] Flanagan L, Schmid J, Ebert M, Soucek P, Kunicka T, Liska V, Bruha J, Neary P, Dezeeuw N, Tommasino M, Jenab M, Prehn JH, Hughes DJ. Fusobacterium nucleatum associates with stages of colorectal neoplasia development, colorectal cancer and disease outcome. Eur J Clin Microbiol Infect Dis. 2014 Aug;33(8):1381-90. doi: 10.1007/s10096-014-2081-3. Epub 2014 Mar 6. PMID 24599709
- [Background] Amitay EL, Werner S, Vital M, Pieper DH, Hofler D, Gierse IJ, Butt J, Balavarca Y, Cuk K, Brenner H. Fusobacterium and colorectal cancer: causal factor or passenger? Results from a large colorectal cancer screening study. Carcinogenesis. 2017 Aug 1;38(8):781-788. doi: 10.1093/carcin/bgx053. PMID 28582482
- [Background] Liang JQ, Li T, Nakatsu G, Chen YX, Yau TO, Chu E, Wong S, Szeto CH, Ng SC, Chan FKL, Fang JY, Sung JJY, Yu J. A novel faecal Lachnoclostridium marker for the non-invasive diagnosis of colorectal adenoma and cancer. Gut. 2020 Jul;69(7):1248-1257. doi: 10.1136/gutjnl-2019-318532. Epub 2019 Nov 27. PMID 31776231
- [Background] Heitman SJ, Ronksley PE, Hilsden RJ, Manns BJ, Rostom A, Hemmelgarn BR. Prevalence of adenomas and colorectal cancer in average risk individuals: a systematic review and meta-analysis. Clin Gastroenterol Hepatol. 2009 Dec;7(12):1272-8. doi: 10.1016/j.cgh.2009.05.032. Epub 2009 Jun 10. PMID 19523536
- [Background] Yamaji Y, Mitsushima T, Ikuma H, Watabe H, Okamoto M, Kawabe T, Wada R, Doi H, Omata M. Incidence and recurrence rates of colorectal adenomas estimated by annually repeated colonoscopies on asymptomatic Japanese. Gut. 2004 Apr;53(4):568-72. doi: 10.1136/gut.2003.026112. PMID 15016753
- [Background] Robertson DJ, Lee JK, Boland CR, Dominitz JA, Giardiello FM, Johnson DA, Kaltenbach T, Lieberman D, Levin TR, Rex DK. Recommendations on Fecal Immunochemical Testing to Screen for Colorectal Neoplasia: A Consensus Statement by the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2017 Apr;152(5):1217-1237.e3. doi: 10.1053/j.gastro.2016.08.053. Epub 2016 Oct 19. PMID 27769517
- [Background] Hassan C, Antonelli G, Dumonceau JM, Regula J, Bretthauer M, Chaussade S, Dekker E, Ferlitsch M, Gimeno-Garcia A, Jover R, Kalager M, Pellise M, Pox C, Ricciardiello L, Rutter M, Helsingen LM, Bleijenberg A, Senore C, van Hooft JE, Dinis-Ribeiro M, Quintero E. Post-polypectomy colonoscopy surveillance: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2020. Endoscopy. 2020 Aug;52(8):687-700. doi: 10.1055/a-1185-3109. Epub 2020 Jun 22. PMID 32572858
- [Background] Lee JK, Liles EG, Bent S, Levin TR, Corley DA. Accuracy of fecal immunochemical tests for colorectal cancer: systematic review and meta-analysis. Ann Intern Med. 2014 Feb 4;160(3):171. doi: 10.7326/M13-1484. PMID 24658694